CLINICAL TRIAL: NCT06445374
Title: A Phase 1b Open-Label Exploratory Study Evaluating Inhaled Epinephrine in Individuals With Known or Suspected Metabisulfite Sensitivity Experiencing Systemic Allergic Reactions During Allergy Testing Immunotherapy or Oral Challenges
Brief Title: Effects of Inhaled Epinephrine on Systemic Allergic Reactions During Allergy Testing Immunotherapy or Oral Challenges
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. George Luciuk (Other)
Responsible Party: Sponsor-Investigator, Dr. George Luciuk, Founder, Chief Medical Officer, Kokua Pharma Inc.
Organization: Kokua Pharma Inc. (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GHL-101
Record Dates: First submitted 2024-05-30; First posted 2024-06-06 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Hypersensitivity; Anaphylaxis
Keywords: Immunotherapy; Epinephrine; Upper airway laryngeal edema; Upper airway pharyngeal edema; Hypersensitivity; Hypersensitivity, immediate; Anaphylaxis; Vasoconstrictor agents; Adrenergic alpha-Agonists; Adrenergic beta-Agonists; Bronchodilator agents
MeSH Terms: conditions — Hypersensitivity; Anaphylaxis; Hypersensitivity, Immediate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Inhaled Epinephrine (Experimental): The first inhalation will be administered as soon as possible (i.e., within approximately 30 seconds) following identification of a Grade 2 or greater SAR and confirmation of enrollment by the Principal Investigator. The second inhalation will be administered approximately 10 seconds later, and the subject will be observed for approximately 2 minutes for signs of symptom resolution.
  Inhalations will continue in this manner until either:
  1. resolution of systemic symptoms (defined as a reduction in SAR Grade to ≤1), or
  2. maximum number of inhalations (8 inhalations) is reached, or
  3. administration of intra-muscular epinephrine, whichever occurs earlier
  Interventions: Drug: Inhaled Epinephrine

INTERVENTIONS:
Drug: Inhaled Epinephrine — 0.125 mg per inhalation.
  The maximum proposed dose to be administered is 1.0 mg (consisting of 8 inhalations of 0.125 mg over 6 minutes).

SUMMARY:
The purpose of this exploratory study is to evaluate the effects of inhaled epinephrine in patients with known or suspected metabisulfite sensitivity who experience a systemic allergic reaction (SAR) while undergoing allergy testing, immunotherapy or oral challenges.

DETAILED DESCRIPTION:
This is a Phase 1b, single-center, open label exploratory study that will evaluate the effects of inhaled epinephrine in patients with known or suspected metabisulfite sensitivity and who are undergoing planned allergy testing, subcutaneous immunotherapy (SCIT), oral challenges (food and/or drug), or oral immunotherapy (OIT). This study will enroll and dose up to 60 patients.

The maximum duration of subject participation is approximately 1 week.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, aged ≥ 18 years with known or suspected metabisulfite sensitivity who can also have a clinical history of immunoglobulin E (IgE)-mediated allergy, including a documented sensitivity to allergens (i.e., positive skin prick test, or positive in vitro serum IgE).
2. Have undergone either a) allergy testing for suspected sensitivity/allergy, b) oral challenge (food and/or drug), c) oral immunotherapy (OIT) to treat existing allergies or d) subcutaneous immunotherapy (SCIT) following a prior allergic reaction AND experiences a systemic allergic reaction (SAR) rated as Grade ≥2, following allergy testing, SCIT, oral challenge (food and/or drug), or OIT, and deemed eligible for enrollment by the Principal Investigator.
3. For females of child-bearing potential, not pregnant or lactating, willing to use a highly effective method of birth control between Screening and End-of-Study Visits.

Exclusion Criteria:

1. Known reaction or sensitivity to epinephrine or any of the ingredients of inhaled epinephrine.
2. Known history or presence of clinically relevant cardiovascular, respiratory, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, psychological or other disease/condition that could confound the results of the study or place the subject at undue or additional risk per the judgment of the Investigator.
3. Uncontrolled asthma or chronic obstructive pulmonary disease (COPD).
4. Recent life-threatening asthma within the last 6 months which required admission to hospital prior to study start.
5. Use of any tobacco or of any inhaled products, including vaping and water pipes (Hookahs) within 12 months prior to screening and/or a 10 pack per year history of use.
6. Use of antihistamines within 5 days and/or bronchodilators within 24 hours of pre-challenge visit.
7. Surgical procedures within 90 days of screening that could result in confounding of results or additional risk to the subject, per the judgment of the Investigator.
8. Abnormal vital signs at screening (i.e., systolic blood pressure: < 90 or >140 mmHg, diastolic blood pressure: < 40 or > 90 mmHg or, Heart rate: < 45 or > 100 bpm), respiration rate < 8 or > 20 resp./min.
9. Females who are pregnant, plan to become pregnant or lactating.
10. Participation in another clinical study involving an investigational drug within 30 days prior to screening, an investigational biologic within 60 days prior to screening, or current/planned participation in another interventional study during this study.
11. Previous treatment in this study.
12. Any other reason that, in the opinion of the Investigator, is likely to unfavourably alter subject risk-benefit, confound results, or make it difficult for the subject to fully comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Time to resolution of systemic symptoms. | From first dose administration to 60 minutes following first dose administration.
  Defined as a reduction in systemic allergic reaction (SAR) Grade to ≤ 1.

CONTACTS AND LOCATIONS:
Overall Officials: George H. Luciuk, MD, Principal Investigator — Kokua Pharma Inc.
Locations (1):
- 1232176 Bc Ltd, Richmond, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected during the trial, after deidentification
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Immediately after publication, and for a period of 5 years.
Access Criteria: Any purpose. URL to be added.